CLINICAL TRIAL: NCT02980965
Title: A Randomized Controlled Study to Evaluate the Efficacy and Safety of Endocrine Therapy Plus Chemotherapy Versus Chemotherapy Alone as the Neoadjuvant Therapy in the Treatment of ER-positive, HER2-negative Breast Cancer (IIa-IIIc)
Brief Title: Neoadjuvant Chemo-endocrine Therapy Versus Chemotherapy Alone in ER-positive, HER2-negative Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Director of Department of Surgical Oncology,Cancer Hospital & Institute, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCET-trial
Record Dates: First submitted 2016-11-26; First posted 2016-12-02 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Breast Cancer Female
Keywords: breast cancer; neoadjuvant chemotherapy; endocrine therapy; concurrent
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; Leuprolide; Fluorouracil; Epirubicin; Cyclophosphamide; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- neoadjuvant chemo-endocrine therapy (Experimental): In the experimental arm, patients received concurrent chemotherapy (fluorouracil 500mg/m2 IV, epirubicin 90mg/m2 IV and cyclophosphamide 500mg/m2 IV on day 1 at 3-weekly intervals for 3 cycles followed by docetaxel 100mg/m2 IV on day 1 at 3-weekly intervals for 3 cycles; or epirubicin 90mg/m2 IV and cyclophosphamide 600mg/m2 IV on day 1 at 2-weekly intervals for 4 cycles, followed by docetaxel 100mg/m2 IV on day 1 at 2-weekly intervals for 4 cycles) with endocrine therapy (letrozole with or without leuprorelin) as a neoadjuvant treatment
  Interventions: Drug: letrozole, leuprorelin, fluorouracil, epirubicin, cyclophosphamide, docetaxel
- neoadjuvant chemotherapy alone (Active Comparator): In the control group, patients received neoadjuvant chemotherapy alone (fluorouracil 500mg/m2 IV, epirubicin 90mg/m2 IV and cyclophosphamide 500mg/m2 IV on day 1 at 3-weekly intervals for 3 cycles followed by docetaxel 100mg/m2 IV on day 1 at 3-weekly intervals for 3 cycles; or epirubicin 90mg/m2 IV and cyclophosphamide 600mg/m2 IV on day 1 at 2-weekly intervals for 4 cycles, followed by docetaxel 100mg/m2 IV on day 1 at 2-weekly intervals for 4 cycles)
  Interventions: Drug: fluorouracil, epirubicin, cyclophosphamide, docetaxel

INTERVENTIONS:
Drug: letrozole, leuprorelin, fluorouracil, epirubicin, cyclophosphamide, docetaxel — Postmenopausal patients were treated with letrozole 2.5mg/day p.o until complement of neoadjuvant chemotherapy before surgery, while premenopausal ones received letrozole 2.5mg/day p.o and a subcutaneous injection of the GnRH-a, leuprorelin, as concomitant treatment with neoadjuvant chemotherapy (fluorouracil 600mg/m2 IV, epirubicin 90mg/m2 IV and cyclophosphamide 600mg/m2 IV on day 1 at 3-weekly intervals for 3 cycles followed by docetaxel 100mg/m2 IV on day 1 at 3-weekly intervals for 3 cycles; or epirubicin 90mg/m2 IV and cyclophosphamide 600mg/m2 IV on day 1 at 2-weekly intervals for 4 cycles, followed by docetaxel 80mg/m2 IV on day 1 at 2-weekly intervals for 4 cycles), letrozole was delivered after 1 week of first dose of leuprorelin injection.
  Other Names: GnRH-a, ENANTONE
  Arms: neoadjuvant chemo-endocrine therapy
Drug: fluorouracil, epirubicin, cyclophosphamide, docetaxel — Patients received fluorouracil 500mg/m2 IV, epirubicin 90mg/m2 IV and cyclophosphamide 500mg/m2 IV on day 1 at 3-weekly intervals for 3 cycles followed by docetaxel 100mg/m2 IV on day 1 at 3-weekly intervals for 3 cycles; or epirubicin 90mg/m2 IV and cyclophosphamide 600mg/m2 IV on day 1 at 2-weekly intervals for 4 cycles, followed by docetaxel 100mg/m2 IV on day 1 at 2-weekly intervals for 4 cycles.
  Arms: neoadjuvant chemotherapy alone

SUMMARY:
This was an open-label, randomized controlled trial that aims to compare the efficacy and safety of the concurrent neoadjuvant chemotherapy with endocrine therapy and neoadjuvant chemotherapy alone in ER-positive, HER2-negative breast cancer.

DETAILED DESCRIPTION:
Data showed that concurrent neoadjuvant chemotherapy with endocrine therapy was a effective option for ER-positive, HER2-negative breast cancer patients. However this is still a controversial issue. The present study is an open-label randomized controlled clinical trial that aims to investigate the efficacy of concurrent NCT with endocrine therapy (AI with or without GnRH-a) in patients with ER-positive, HER2-negative breast carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Estrogen receptor-positive and HER2-negative breast cancer patients, with histological stage of IIa-IIIc.
2. Without previous chemotherapy or endocrine therapy.
3. ECOG scores of 0-2 points
4. With measurable and evaluable breast tumor pathologically confirmed as invasive ductal carcinoma
5. Age: 18-70 years
6. Lateral breast cancer
7. Normal or acceptable kidney, liver, cardiovascular, and bone marrow functions

Exclusion Criteria:

1. Pregnant women or nursing mothers
2. With distant metastasis
3. With a history of malignant tumor or complicated with other malignant tumors in addition to breast cancer, except for non-melanoma skin cancer, in situ cervical cancer or other cured malignant tumor without the basis of recurrence for at least five years
4. With mental illness or other conditions affecting the patient compliance
5. With other serious diseases or medical conditions:

   1. Congestive heart failure or unstable angina pectoris, myocardial infarction within 6 months before the enrollment, uncontrolled hypertension and uncontrolled high-risk arrhythmia considered by the investigator
   2. Obvious neurological or psychiatric disorders, including psychosis, epileptic dementia and other diseases may affect the understanding and sign of the informed consent for
   3. Uncontrolled acute infection
6. Concurrent use of other investigational drugs; or participating in other clinical trials involving investigational drugs within 30 days before this study
7. With allergic constitution and any known or suspected drug allergy
8. Not suitable for the trial considered by the investigator

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2013-05; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
objective response rate (ORR) | 4 years
  the proportion of patients achieving clinical complete response and partial response in the breast based on magnetic resonance imaging

SECONDARY OUTCOMES:
Ki67 proliferation marker changes | 4 years
  Absolute Ki67 change as well as geometric mean percentage change in Ki67 positivity
pathologic complete response (pCR) | 4 years
  Disappearance of residual invasive disease (residual ductal carcinoma in situ allowed) in breast and the absence of positive lymph nodes
pathological response rate | 4 years
  The proportion of patients achieving pathological response based on Miller-Payne grading system
Progression-free survival (DFS) | 6 years
  The interval between the date of randomization to disease progression during treatment, any recurrence, contralateral breast cancer, the appearance of a second primary cancer, or death not due to cancer, whichever occurred first.
Incidence of Serious Treatment-Emergent Adverse Events(grade 3 or 4) | 4 years
  Assessed according to National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Min Shao, MD, Principal Investigator — Cancer Hospital/ Institute, Fudan University
Locations (1):
- Cancer Hospital/ Institute, Fudan University, Shanghai, Shanghai Municipality, China